CLINICAL TRIAL: NCT04352413
Title: An Open-label, Multi-center, Phase 2 Study of Liposome-entrapped Mitoxantrone Hydrochloride Injection (PLM60) in Subjects With Relapsed Small-cell Lung Cancer After Platinum-based First-Line Chemotherapy
Brief Title: A Study of PLM60 in Subjects With Relapsed Small-cell Lung Cancer After Platinum-based First-Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-010
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2020-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: PLM60 (Experimental): 20 mg/m2, 4 weeks/cycle, administered on day 1 of each cycle
  Interventions: Drug: PLM60
- Cohort B: PLM60 (Experimental): 15mg/m2, 3 weeks/cycle, administered on day 1 of each cycle
  Interventions: Drug: PLM60

INTERVENTIONS:
Drug: PLM60 — Administration: Intravenous infusion

SUMMARY:
This is an open, multicenter phase II clinical study for PLM60. The primary aim of the study is to observe the initial efficacy of PLM60 in treatment of small cell lung cancer. The secondary aim is to explore the safety and PK characteristics of PLM60

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of SCLC;
2. Must have recurrence or progression after platinum-based first-line chemotherapy or chemoradiation therapy for the treatment of SCLC;
3. ECOG performance status 0~2;
4. Measurable lesion according to RECIST v1.1;
5. Life expectancy ≥ 12 weeks;
6. Adequate organ function;
7. Signed informed consent from the patient.

Exclusion Criteria:

1. Radical surgical treatment for primary small cell lung cancer;
2. Any anti-tumor treatment received within 4 weeks before the first use of the study drug;
3. Untreated or symptomatic central nervous system (CNS) metastases;
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
5. History of serious systemic diseases;
6. History of serious autoimmune diseases;
7. Those receiving treatment of adriamycin or other anthracyclines previously, with the total cumulative adriamycin (or adriamycin-equivalent) dose of >360 mg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 2 year
  To evaluate ORR in SCLC subjects treated with PLM60

SECONDARY OUTCOMES:
Duration of Response (DoR) | Through study completion, an average of 2 year
  To evaluate DoR in SCLC subjects treated with PLM60
Disease Control Rate (DCR) | Through study completion, an average of 2 year
  To evaluate DCR in SCLC subjects treated with PLM60
Progression Free Survival (PFS) | Through study completion, an average of 2 year
  To evaluate PFS in SCLC subjects treated with PLM60
Overall Survival (OS) | Through study completion, an average of 2 year
  To evaluate OS in SCLC subjects treated with PLM60
Adverse Events | Through study completion, an average of 2 year
  To evaluate the safety profiles in SCLC subjects treated with PLM60
Serious Adverse Events (SAEs) | Through study completion, an average of 2 year
  To evaluate the safety profiles in SCLC subjects treated with PLM60

CONTACTS AND LOCATIONS:
Overall Officials: Kun Lou, Study Chair — Department of Medicine, CSPC Clinical Development Division
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No